CLINICAL TRIAL: NCT07276217
Title: Phacoemulsification and Intraocular Lens Implantation: Patient Registry
Status: Recruiting | Type: Observational
Sponsor: Sensor Cliniq (Other)
Responsible Party: Principal Investigator, Jakub Polinski, Ophthalmologist, Medical Doctor, Sensor Cliniq
Other Study IDs: KB/1520/24
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Cataract; Intraocular Lens
Keywords: cataract; intraocular lens; phacoemulsification
MeSH Terms: conditions — Cataract | interventions — Lenses, Intraocular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Bilateral Monofocal IOL: Patients who underwent bilateral cataract surgery with implantation of monofocal intraocular lenses in both eyes between 2021 and 2025, and attended a follow-up visit.
  Interventions: Device: Intraocular lens
- Bilateral Monofocal-plus IOL: Patients who underwent bilateral cataract surgery with implantation of monofocal-plus intraocular lenses in both eyes between 2021 and 2025, and attended a follow-up visit.
  Interventions: Device: Intraocular lens
- Bilateral EDOF IOL: Patients who underwent bilateral cataract surgery with implantation of extended-depth-of-focus (EDOF) intraocular lenses in both eyes between 2021 and 2025, and attended a follow-up visit.
  Interventions: Device: Intraocular lens

INTERVENTIONS:
Device: Intraocular lens — Implantation of an intraocular lens following phacoemulsification cataract extraction, with lens type selected according to routine clinical practice (e.g., monofocal, toric, multifocal, or extended-depth-of-focus).

SUMMARY:
The aim of the study is to create a patient registry that will allow for comparison of cataract treatment outcomes using phacoemulsification with implantation of different types of intraocular lenses.

DETAILED DESCRIPTION:
This study will establish a registry to evaluate outcomes associated with intraocular lens implants in patients undergoing cataract surgery. Retrospective assessments will include routinely collected preoperative, intraoperative, and postoperative data. Prospectively, visual acuity, refraction, examination findings, patient-reported outcomes, and complications will be collected for up to 60 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone cataract surgery or are scheduled for bilateral cataract surgery with implantation of an extended-depth-of-focus (EDOF) intraocular lens, a monofocal-plus intraocular lens, or a standard monofocal intraocular lens.

Exclusion Criteria:

* Anterior or posterior segment pathologies affecting postoperative visual acuity, including but not limited to: severe dry eye syndrome, corneal dystrophies, uveitis, retinal degenerative changes, glaucoma, or diabetic retinopathy.
* Pseudoexfoliation syndrome
* Keratoconus
* History of laser refractive surgery
* Prior ocular surgery other than cataract surgery
* Amblyopia
* Posterior capsule opacification
* Postoperative best-corrected visual acuity (BCVA) less 0.5
* Intraoperative complications, including posterior capsule rupture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone or are scheduled for bilateral cataract surgery at Sensor Cliniq between 2021 and 2025.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Corrected and Uncorrected Distance, Intermediate and Near Visual Acuity | Measured at the follow-up visit up to 60 months after cataract surgery
  Distance, intermediate, and near visual acuity will be measured both uncorrected and corrected using standard ETDRS charts at 4 meters for distance, 66 cm for intermediate, and 40 cm for near visual acuity.

SECONDARY OUTCOMES:
Objective Refraction | Measured at the follow-up visit up to 60 months after cataract surgery
  Spherical and cylindrical refractive errors will be measured objectively using an autorefractometer.
Subjective Refraction | Measured at the follow-up visit up to 60 months after cataract surgery
  Spherical and cylindrical refractive errors will be measured subjectively using trial frame glasses and patient responses.
Monocular and Binocular Defocus Curve | Measured at the follow-up visit up to 60 months after cataract surgery
  Visual acuity will be measured at varying defocus levels under monocular and binocular conditions to assess the range of functional vision. Measurements will be taken in 0.5 D steps from +1.00 D to -2.50 D.
Contrast Sensitivity | Measured at the follow-up visit up to 60 months after cataract surgery
  Contrast sensitivity will be assessed using the Matrix Perceptix test under photopic light conditions.
Keratometry | Measured at the follow-up visit up to 60 months after cataract surgery
  Keratometry will be measured using IOLMaster 500 and Pentacam
Anterior Chamber Depth | Measured at the follow-up visit up to 60 months after cataract surgery
  Anterior chamber depth will be measured using IOLMaster 500 and Pentacam.
Pupil Size | Measured at the follow-up visit up to 60 months after cataract surgery
  Pupil diameter will be measured using IOLMaster 500 and Pentacam.
Central Corneal Thickness | Measured at the follow-up visit up to 60 months after cataract surgery
  Central corneal thickness will be measured using Pentacam.
Anterior Chamber Angle | Measured at the follow-up visit up to 60 months after cataract surgery
  Anterior chamber angle will be measured using Pentacam.
Primary and Secondary Spherical Aberrations | Measured at the follow-up visit up to 60 months after cataract surgery
  Primary and secondary spherical aberrations will be measured using Pentacam.
Patient-Reported Spectacle Independence | Measured at the follow-up visit up to 60 months after cataract surgery
  Degree of spectacle independence will be assessed using the Patient-Reported Spectacle Independence Questionnaire (PRSIQ).
Patient-Reported Quality of Vision | Measured at the follow-up visit up to 60 months after cataract surgery
  Quality of vision will be assessed using the Quality of Vision Questionnaire (QoV).

CONTACTS AND LOCATIONS:
Locations (1):
- Sensor Cliniq, Warsaw, Poland